CLINICAL TRIAL: NCT00234442
Title: A Phase II, Multicentre, Non-Comparative, Open-Label Study To Evaluate The Efficacy And Tolerability Of ZD1839 (Iressa™) In Asymptomatic Radio-Naive Patients With Brain Metastases From Non-Small Cell Lung Carcinoma (NSCLC) Who Have Relapsed Following Prior Chemotherapy
Brief Title: Iressa in the Treatment of Brain Metastases From Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to insufficient recruitment.
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0569
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Brain Neoplasms; Non Small Cell Lung Cancer
Keywords: Non symptomatic brain metastases; Iressa
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

INTERVENTIONS:
Drug: Iressa (Gefitinib)

SUMMARY:
The aim of the study is to determine if Iressa is effective in the treatment of Brain metastases from NCSLC

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed brain metastases from Non Small Cell Lung Cancer
* No symptoms due to brain metastases
* No previous radiotherapy treatment for the Brain metastases

Exclusion Criteria:

* No prior chemotherapy
* No other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47
Dates: Start 2004-07; Study Completion 2006-02

PRIMARY OUTCOMES:
Disease control rate (complete response, partial response and stable disease)

SECONDARY OUTCOMES:
Duration of response
Time to progression
Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Crino, MD, Principal Investigator — Bologna, Italy
Locations (4):
- Italy (4):
  - Research Site, Bologna
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Rozzano